CLINICAL TRIAL: NCT04092036
Title: Prospective Study: Optic Nerve Sheath Diameter in Prediction of Fluid Responsiveness
Brief Title: Optic Nerve Sheath Diameter in Prediction of Fluid Responsiveness
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hadeel Ibraheim Elsagheir, Resident at Anesthesiology, Surgical ICU and Pain Medicine Department, Tanta University
Other Study IDs: 33157/06/19
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Fluid Responsiveness; Optic Nerve Sheath Diameter; Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unstable patients: Patients on mechanical ventilation, 18 years or older and developing hypotension (Mean arterial blood pressure) <65 mmHg
  Interventions: Device: Optic Nerve Sheath Diameter (ONSD) measurement by ultrasound

INTERVENTIONS:
Device: Optic Nerve Sheath Diameter (ONSD) measurement by ultrasound — ONSD measurements will be performed in the supine patient. Ultrasound gel will be applied over the closed upper eyelid. The ultrasound probe will be placed on the temporal area of the eyelid. Then the probe will be angled in order to display the entry of the optic nerve into the globe.
  ONSD will be measured 3 mm behind the globe in the transverse plane perpendicular to the optic nerve. For each optic nerve three measurements will be made. The ONSD corresponds to the mean of the six values which will be obtained from each patient (three measurements for each eye).

SUMMARY:
The aim of the study to examine Optic Nerve Sheath Diameter measurement for prediction of fluid responsiveness in hemodynamically unstable patients

ELIGIBILITY:
Inclusion Criteria:

* Patients on mechanical ventilation
* 18 years or older
* patients developing hypotension (Mean arterial blood pressure) <65 mmHg

Exclusion Criteria:

* Patients with Spontaneously breathing activity.
* Patients with a history of intracranial disease e.g. (stroke, TBI, causes of increased intracranial pressure).
* local cause in the eye as (Glaucoma, Single eye)
* Need for high PEEP.
* Known history of cardiac disease.
* Organ/s failure at admission

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Tanta University Hospitals at the surgical intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2020-03-14 (Estimated); Study Completion 2020-03-14 (Estimated)

PRIMARY OUTCOMES:
The cut-off value of optic nerve sheath diameter (ONSD) for prediction of fluid responsiveness | first day

SECONDARY OUTCOMES:
Correlation between Stroke Volume Variation (by electrical cardiometry) and ONSD | first day

IPD SHARING:
Plan to Share IPD: Yes